CLINICAL TRIAL: NCT07075562
Title: Effects of Transcatheter Hepatic Arterial Chemoembolization (TACE) and Bevacizumab Arterial Perfusion on Tumor Load and Angiogenesis in Patients With Hepatocellular Carcinoma Invading Portal Vein
Brief Title: TACE Plus Bevacizumab for Hepatocellular Carcinoma With Portal Vein Invasion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Bingzheng Yan, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220685
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Observation Group (TACE + Bevacizumab) (Experimental): Patients randomized to this arm received transcatheter hepatic artery chemoembolization (TACE) combined with arterial infusion of bevacizumab.
  Interventions: Drug: Bevacizumab Arterial Perfusion plus TACE
- Active Comparator: Control Group (Conventional Therapy) (Active Comparator): Patients randomized to this arm received conventional therapy for HCC with portal vein invasion, serving as the active control.
  Interventions: Procedure: Conventional Therapy

INTERVENTIONS:
Drug: Bevacizumab Arterial Perfusion plus TACE — The intervention consists of a combination treatment. Patients undergo transcatheter hepatic artery chemoembolization (TACE), a procedure involving localized delivery of chemotherapy and embolization of the tumor-feeding arteries. This is combined with a targeted arterial perfusion of bevacizumab, a monoclonal antibody that inhibits vascular endothelial growth factor (VEGF).
  Arms: Experimental: Observation Group (TACE + Bevacizumab)
Procedure: Conventional Therapy — Patients in the control group received conventional therapy, which typically consists of TACE alone for this patient population. This involves the selective catheterization of hepatic arteries supplying the tumor, followed by the infusion of chemotherapeutic agents and an embolic agent to induce tumor necrosis.
  Arms: Active Comparator: Control Group (Conventional Therapy)

SUMMARY:
This is a prospective, randomized study designed to compare the efficacy of transcatheter hepatic artery chemoembolization (TACE) combined with bevacizumab arterial perfusion versus conventional therapy in patients with hepatocellular carcinoma (HCC) invading the portal vein. The study aims to evaluate the effects on tumor load, angiogenesis, and survival outcomes.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) with portal vein invasion has a poor prognosis and limited therapeutic options. Transcatheter hepatic artery chemoembolization (TACE) is a standard locoregional therapy, but its efficacy can be limited by hypoxia-induced angiogenesis. Bevacizumab, a VEGF inhibitor, can counteract this angiogenic rebound. This study was designed to investigate the potential synergistic effects of combining TACE with bevacizumab arterial perfusion. A total of 180 patients with portal vein-invasive HCC were prospectively recruited and randomized to either the combination therapy group or a conventional therapy control group. The primary objectives were to assess changes in tumor load (size and number), serum angiogenic factors (VEGF and PDGF), and tumor vascular density. Secondary objectives included evaluating safety and comparing progression-free and overall survival between the two groups to establish an evidence-based framework for this treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years.
* Confirmed diagnosis of Hepatocellular Carcinoma (HCC) with radiological evidence of portal vein invasion.
* Preserved liver function (Child-Pugh class A or B).
* Absence of severe cardiac, renal, or other vital organ dysfunctions.
* Complete clinical and follow-up data available.
* Provided written informed consent.

Exclusion Criteria:

* History of other malignancies within the past five years.
* Prior or planned liver transplantation.
* Severe comorbidities (e.g., decompensated cirrhosis, active bleeding, or cardiac disease).
* Pregnant or lactating women.
* Known hypersensitivity to bevacizumab or other components of the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Tumor Load | Baseline (before treatment) and 3 months post-treatmen
  Measured by assessing the change in tumor diameter (in cm) and the total number of tumors from baseline. Measurements are performed using Magnetic Resonance Imaging (MRI).
Change in Serum Angiogenic Factors | Baseline (before treatment) and at the 3-month post-treatment follow-up
  Measured by the change in serum levels of Vascular Endothelial Growth Factor (VEGF) and Platelet-Derived Growth Factor (PDGF) in pg/mL, as quantified by Enzyme-Linked Immunosorbent Assay (ELISA).
Change in Tumor Vascular Density | Baseline (before treatment) and 3 months post-treatment
  Measured as the change in the density of blood vessels (vessels/cm²) in the tumor area, evaluated by Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI).

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until death, with a median follow-up of 24 months (range 12-36 months)
  Time from randomization to death from any cause. Reported as median survival in months.
Progression-Free Survival (PFS) | From date of randomization until disease progression or death, assessed at 6-month intervals up to 36 months
  Time from randomization to disease progression or death from any cause, whichever occurs first. Reported as median survival in months.
Incidence of Adverse Events | From the start of the first intervention until the 3-month post-treatment follow-up visit
  Number and percentage of participants experiencing treatment-related adverse events, graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China